

#### STATISTICAL ANALYSIS PLAN

**Study Title:** A Phase 1 Study to Evaluate the Safety, Tolerability,

Pharmacokinetics, and Pharmacodynamics of GS-5829 as a Monotherapy in Subjects with Advanced Solid Tumors and Lymphomas and in Combination with Exemestane or Fulvestrant

in Subjects with Estrogen Receptor Positive Breast Cancer

Name of Test Drug: GS-5829

Study Number: GS-US-350-1599

**Protocol Version (Date):** Amendment 6 (20 June 2016)

**Analysis Type:** Final Analysis

**Analysis Plan Version:** 1.0

**Analysis Plan Date:** 03 January 2018

Analysis Plan Author(s): PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

# TABLE OF CONTENTS

| STA | ATISTI | CAL ANALYSIS PLAN | 1 |
|---|---|---|---|
| TA | BLE OI | F CONTENTS | 2 |
| LIS | T OF T | ABLES | 3 |
| | | COKINETIC ABBREVIATIONS | |
| 1. | INTRODUCTION | | |
| | 1.1. | Study Objectives | |
| | 1.2. | Study Design | |
| | 1.3. | Sample Size and Power | 10 |
| 2. | TYPE OF PLANNED ANALYSIS | | |
| | 2.1. | Interim Analyses | |
| | 2.2. | Final Analysis | 11 |
| 3. | GEN | ERAL CONSIDERATIONS FOR DATA ANALYSES | 12 |
| | 3.1. | Analysis Sets | 12 |
| | | 3.1.1. All Enrolled Analysis Set | |
| | | 3.1.2. Full Analysis Set | |
| | | 3.1.3. Pharmacokinetic Analysis Set | |
| | 3.2. | Subject Grouping | |
| | 3.3. | Strata and Covariates | |
| | 3.4. Examination of Subject Subgroups | | |
| | 3.5. Multiple Comparisons | | |
| | 3.6. | Missing Data and Outliers | |
| | | 3.6.1. Missing Data | |
| | 2.7 | 3.6.2. Outliers | |
| | 3.7. | Data Handling Conventions and Transformations | |
| | 3.8. | Analysis Visit Windows | |
| | | 3.8.1. Definition of Study Day | |
| | | 3.8.2. Analysis Visit Windows | 13 |
| | | Window | 15 |
| 4. | CHDI | JECT DISPOSITION | |
| 4. | | | |
| | 4.1. | Subject Enrollment and Disposition | |
| | 4.2. | Extent of Study Drug Exposure and Adherence | |
| | | 4.2.1. Duration of Exposure to Study Drug | |
| | 4.2 | 4.2.2. Adherence to GS-5829 | |
| | 4.3. | Protocol Deviations | |
| 5. | BASI | ELINE CHARACTERISTICS | 18 |
| | 5.1. | Demographics | 18 |
| | 5.2. | | |
| | 5.3. | Medical History | |
| | 5.4. | Prior Anticancer Therapy | 18 |
| 6. | EFFI | CACY ANALYSES | 20 |
| | 6.1. Efficacy Endpoint | | |
| | | 6.1.1. Definition of Efficacy Endpoints | |
| | | 6.1.2. Analysis Methods for Efficacy Endpoints | |

| 7. | SAFE | ETY ANA | ALYSES | 22 |
|---|---|---|---|---|
| | 7.1. Adverse Events and Deaths | | se Events and Deaths | 22 |
| | | 7.1.1. | Adverse Event Dictionary | 22 |
| | | 7.1.2. | Adverse Event Severity | 22 |
| | | 7.1.3. | Relationship of Adverse Events to Study Drug | 22 |
| | | 7.1.4. | Serious Adverse Events | |
| | | 7.1.5. | Treatment-Emergent Adverse Events | |
| | | 7.1.6. | Summaries of Adverse Events and Deaths | 23 |
| | | 7.1.7. | Additional Analysis of Adverse Events | 25 |
| | 7.2. | Labora | atory Evaluations | 25 |
| | | 7.2.1. | Summaries of Numeric Laboratory Results | 25 |
| | | 7.2.2. | Graded Laboratory Values | 26 |
| | | 7.2.3. | Liver-related Laboratory Evaluations | 27 |
| | | 7.2.4. | Shifts Relative to the Baseline Value | |
| | 7.3. | Body V | Weight and Vital Signs | 27 |
| | 7.4. | Prior a | and Concomitant Medications | |
| | | 7.4.1. | Prior Medications | |
| | | 7.4.2. | Concomitant Medications | |
| | 7.5. | Electro | ocardiogram Results | |
| | | 7.5.1. | Corrected QT Intervals | |
| | | 7.5.2. | | |
| | 7.6. | | Safety Measures | |
| | 7.7. | Change | es From Protocol-Specified Safety Analyses | 30 |
| 8. | PHARMACOKINETIC (PK) ANALYSES | | | 31 |
| | 8.1. | 8.1. PK Sample Collection | | 31 |
| | | 8.1.1. | Estimation of PK Parameters | 31 |
| | | 8.1.2. | PK Parameters | 31 |
| 9. | REFE | ERENCES | S | 34 |
| 10. | SOFT | WARE | | 35 |
| 11. | SAP 1 | REVISIO | )N | 36 |
| 12 | APPF | ENDICES | S | 37 |
| 12. | 71172 | or (Brebs | | |
| | Appendix 1. | | Schedule of Assessments | 37 |
| | Appendix 2. | | List of Medical Search Terms for Decreased Platelets | 41 |
| | Appendix 3. | | List of Medical Search Terms for Haemorrhage | 42 |
| | Appendix 4. | | List of Medical Search Terms for Diarrhoea | 61 |
| | | | LIST OF TABLES | |
| | Table | . 1 | PK Parameters for Analytes | 22 |
| | 1 4010 | | 1 11 1 urumowio 101 / mury wo | |

#### LIST OF ABBREVIATIONS

AE adverse event

AEI adverse event of interest
ALT alanine aminotransferase
AST aspartate aminotransferase
BLQ below the limit of quantitation

BMI body mass index
BOR best overall response
CI confidence interval
CR complete response
CRF case report form
CSR clinical study report

CTCAE Common Toxicity Criteria for Adverse Events

DILI drug-induced liver injury
DLT dose-limiting toxicity
DMC data monitoring committee

ECG electrocardiogram
ET early termination
FAS Full Analysis Set
Hb hemoglobin
HLT high-level term

ICH International Conference on Harmonization (of Technical Requirements for Registration of

Pharmaceuticals for Human Use)

LTT lower-level term
LOQ limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

MTD maximum tolerated dose

NE not evaluable

ORR overall response rate
PD progressive disease
PFS progression-free survival

PK pharmacokinetics
PR partial response
PT preferred term

Q1, Q3 first quartile, third quartile

QRS electrocardiographic deflection between the beginning of the Q wave and termination of the

S wave representing time for ventricular depolarization

QT electrocardiographic interval between the beginning of the Q wave and termination of the T wave

representing the time for both ventricular depolarization and repolarization to occur

QTc QT interval corrected for heart rate

QTcF QT interval corrected for heart rate using Fridericia's formula

RP2D recommended phase 2 dose

RR electrocardiographic interval representing the time measurement between the R wave of one

heartbeat and the R wave of the preceding heartbeat

SAE serious adverse event SAP statistical analysis plan

SD stable disease StD standard deviation

SI (units) international system of units

SOC system organ class

TEAE treatment-emergent adverse event

TFLs tables, figures, and listings
ULN upper limit of normal

VR ventricular rate

WHO World Health Organization

#### PHARMACOKINETIC ABBREVIATIONS

AUC<sub>last</sub> area under the concentration versus time curve from time zero to the last quantifiable concentration

AUC<sub>tau</sub> area under the concentration versus time curve over the dosing interval

C<sub>last</sub> last observed quantifiable concentration of the drug

C<sub>max</sub> maximum observed concentration of drug

C<sub>tau</sub> observed drug concentration at the end of the dosing interval CLss/F apparent oral clearance after administration of the drug:

at steady state: CLss/F = Dose/AUC<sub>tau</sub>, where "Dose" is the dose of the drug

 $t_{1/2}$  estimate of the terminal elimination half-life of the drug, calculated by dividing the natural log of 2

by the terminal elimination rate constant  $(\lambda_z)$ 

 $T_{last}$  time (observed time point) of  $C_{last}$   $T_{max}$  time (observed time point) of  $C_{max}$ 

 $\lambda_{\rm Z}$  terminal elimination rate constant, estimated by linear regression of the terminal elimination phase

of the concentration of drug versus time curve

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the clinical study report (CSR) for Study GS-US-350-1599. This SAP is based on the study protocol amendment 6 dated 20 June 2016 and the electronic case report form (eCRF). The SAP will be finalized before database finalization. Any changes made after the finalization of the SAP will be documented in the CSR.

#### 1.1. Study Objectives

The primary objectives of this study are as follows:

- Characterize the safety and tolerability of GS-5829 as a monotherapy in subjects with advanced solid tumors and lymphomas
- Determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of GS-5829 as a monotherapy in subjects with advanced solid tumors and lymphomas
- Characterize the safety and tolerability of GS-5829 in combination with exemestane or fulvestrant in subjects with advanced estrogen receptor positive breast cancer
- Determine the MTD or RP2D of GS-5829 in combination with exemestane or fulvestrant in subjects with advanced estrogen receptor positive breast cancer

The secondary objective of this study is as follows:

 Evaluate the pharmacokinetics (PK) of GS-5829 alone in subjects with advanced solid tumors and lymphomas and in combination with exemestane or fulvestrant in subjects with advanced estrogen receptor positive breast cancer



## 1.2. Study Design

This is an open-label, multicenter, sequential dose-escalation study to evaluate the safety, tolerability, PK, and PD of GS-5829 as a single agent in subjects with advanced solid tumors and lymphomas and in combination with exemestane or fulvestrant in subjects with advanced estrogen receptor positive breast cancer.

#### Group 1: Single agent GS-5829 in solid tumors and lymphomas

Cohorts of subjects with advanced solid tumors and lymphomas who have failed or are intolerant to standard therapy or for whom no standard therapy exists will be sequentially enrolled at progressively higher dose levels to receive oral GS-5829 as monotherapy once daily (QD). The starting dose will be 0.6 mg. Each dose level will enroll 1 subject until a  $\geq$  Grade 2 treatment related toxicity is observed within the initial dosing period (Study Day 1 through Cycle 1 Day 28 for all cohorts). At Dose Level 5 or if a  $\geq$  Grade 2 treatment related toxicity is observed (whichever occurs first), the dose level will be expanded to 3 subjects. (Note: subjects enrolled with Grade 2 hemoglobin [Hb] must have Hb worsen by at least 1 grade from baseline to be considered for expansion of the cohort to 3 subjects).

Once a dosing level has been expanded to 3 subjects, a standard 3+3 study design will begin and, dose escalation [3+3] will be performed at every subsequent dose level with cohort sizes of 3 to 6 subjects. Subjects in the first 3 cohorts will receive a single dose and then approximately 7 days later, initiate dosing once daily.

The doses for each Dose Level are shown in the table below.

**Group 1: Single Agent GS-5829** 

| Dose Level | GS-5829* |
|------------|----------|
| 1 | 0.6 mg |
| 2 | 1.4 mg |
| 3 | 2 mg |
| 4 | 3 mg |
| 5 | 4 mg |
| 6 | 6 mg |
| 7 | 9 mg |
| 8 | 12 mg |

<sup>\*</sup> Dose Levels may be modified based on emerging safety and PK results.

If a dose limiting toxicity (DLT) occurs within the 28 day DLT period at any dose level, this level will be expanded to enroll 3 additional subjects.

The safety and tolerability of each dose level will be assessed by a safety review team (SRT) after all subjects in the cohort have been followed for at least 28 days after the first dose of GS-5829. If no DLTs occur in up to 3 subjects or < 2 DLTs occur in up to 6 subjects on any dose level after 28 days on treatment, the next dose level will open. Each subsequent dose level will open if the dose level preceding has no DLTs in 3 subjects or < 2 DLTs in up to 6 subjects.

# Group 2: Combination therapy of GS-5829 with exemestane or fulvestrant in patients with advanced stage estrogen receptor positive breast cancer

Cohorts of subjects with advanced stage estrogen receptor positive breast cancer for whom no standard curative therapy exists and who are candidates for exemestane or fulvestrant will be sequentially enrolled at progressively higher dose levels of oral GS-5829 in combination with full standard doses of exemestane or fulvestrant. The starting dose of GS-5829 will be 2.0 mg QD, which is a dose level that has been demonstrated to be safe and tolerable (no Grade 2 or higher drug related toxicity) as a single agent in patients with solid tumors. Dose escalation will continue with cohort sizes of 3-6 subjects in parallel arms: Group 2A will initiate with 2.0 mg of GS-5829 orally once daily on Cycle 1 Day 1 combined with 25 mg of exemestane administered once daily beginning on Cycle 1 Day 1. The subject may initiate exemestane any time prior to, or on, Cycle 1 Day 1. Group 2B will initiate with 2.0 mg of GS-5829 orally once daily on Cycle 1 Day 1 with 500 mg fulvestrant administered intramuscularly Cycle 1 Day 1 and then every 28 days (+/- 3 days). If Cycle 1 Day 1 is the subject's first dose of fulvestrant, a one-time additional dose of fulvestrant should be administered on Cycle 1 Day 15.

The candidate doses of GS-5829 for each Dose Level for Group 2 are shown in the table below.

| <b>Group 2: Combination of G</b> | GS-5829 in Breast Cancer |
|----------------------------------|--------------------------|
|----------------------------------|--------------------------|

| Dose Level | GS-5829* | Group 2A Exemestane | Group 2B Fulvestrant |
|---|---|---|---|
| 1 | 2 mg | | |
| 2 | 3 mg | | |
| 3 | 4 mg | 25 mg amily and daily | 500 mg intramuscularly day 1, 29 |
| 4 | 6 mg | 25 mg orally once daily | and then every 28 days** |
| 5 | 9 mg | | |
| 6 | 12 mg | | |

<sup>\*</sup> Dose Levels may be modified based on emerging safety and PK results.

Group 2A and Group 2B will dose escalate independent of each other. In both Groups 2A and Group 2B, each cohort will consist of 3 newly enrolled subjects who will be treated at the specified dose level. After all subjects in each cohort have been followed for at least 28 days after the first dose of GS-5829, a dose-DLT model (Bayesian logistic regression model) utilizing all available GS-5829 safety data will be built, and will provide estimates of DLT rates at all dose levels.

<sup>\*\*</sup> Subjects initiating fulvestrant on this study should receive a single additional dose of fulvestrant on Cycle 1 Day 15.

# 1.3. Sample Size and Power

The sample size of the study is determined based on the number of dose levels evaluated and the emerging GS-5829-related toxicities. The study will consist of up to 120 subjects.

A total of 33 subjects were enrolled when the study was completed.

# 2. TYPE OF PLANNED ANALYSIS

## 2.1. Interim Analyses

This study does not have a data monitoring committee (DMC). Therefore, no analyses will be conducted for the DMC.

No formal interim efficacy analysis, which may lead to early termination for efficacy or futility, is planned.

# 2.2. Final Analysis

After all subjects have completed the study, outstanding data queries have been resolved or adjudicated as unresolvable, and the data have been cleaned and finalized, the final analysis of the data will be performed.

#### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects (n), mean, standard deviation (StD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

By-subject listings will be presented for all subjects in the All Enrolled Analysis Set and sorted by subject ID number, visit date, and time (if applicable). Data collected on log forms, such as adverse events, will be presented in chronological order within the subject. The study group and dose level to which subjects were initially assigned will be used in the listings. Age, sex at birth, race, and ethnicity will be included in the listings, as space permits.

#### 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. The analysis set will be identified and included as a subtitle of each table, figure, and listing.

For each analysis set, the number and percentage of subjects eligible for inclusion, as well as the number and percentage of subjects who were excluded, will be summarized by study group and dose level.

A listing of reasons for exclusion from analysis sets will be provided by subject.

## 3.1.1. All Enrolled Analysis Set

All Enrolled Analysis Set includes all subjects who received a study subject identification number in the study after screening.

#### 3.1.2. Full Analysis Set

The Full Analysis Set (FAS) includes all subjects who took at least 1 dose of study drug. This is the primary analysis set for efficacy analyses and safety analyses.

#### 3.1.3. Pharmacokinetic Analysis Set

The Pharmacokinetic (PK) Analysis Set will include all enrolled subjects who took at least 1 dose of study drug and have at least 1 nonmissing postdose value reported by the PK laboratory. This is the primary analysis set for all PK analyses.

## 3.2. Subject Grouping

For analyses based on the FAS, subjects will be grouped according to the actual treatment received.

For the PK Analysis Set, subjects will be grouped according to the actual treatment they received.

#### 3.3. Strata and Covariates

This study does not use a stratified randomization schedule when enrolling subjects. No covariates will be included in safety analyses.

## 3.4. Examination of Subject Subgroups

There are no prespecified subject subgroupings for safety analyses.

#### 3.5. Multiple Comparisons

Adjustments for multiplicity will not be made, because no formal statistical testing will be performed in this study.

#### 3.6. Missing Data and Outliers

#### 3.6.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified. Exceptions are presented in this document.

For missing last dosing date of study drug, imputation rules are described in Section 4.2.1. The handling of missing or incomplete dates, for adverse event (AE) onset is described in Section 7.1.5.2, and for prior and concomitant medications in Section 7.4.

#### **3.6.2. Outliers**

Outliers will be identified during the data management and data analysis process, but no sensitivity analyses will be conducted. All data will be included in the data analysis.

## 3.7. Data Handling Conventions and Transformations

In general, age (in years) on the date of the first dose of study drug will be used for analyses and presentation in listings. If an enrolled subject was not dosed with any study drug, the enrollment date will be used instead of the first dosing date of study drug. For screen failures, the date the informed consent was signed will be used for age calculation. If only the birth year is collected on the CRF, "01 July" will be used for the unknown birth day and month for the purpose of age calculation. If only birth year and month are collected, "01" will be used for the unknown birth day.

Non-PK data that are continuous in nature but are less than the lower limit of quantitation (LOQ) or above the upper LOQ will be imputed as follows:

• A value that is 1 unit less than the LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "< x" (where x is considered the LOQ). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used to calculate summary statistics. An exception to this rule is any value reported as < 1 or < 0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used to calculate summary statistics.

- A value that is 1 unit above the LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "> x" (where x is considered the LOQ). Values with decimal points will follow the same logic as above.
- The LOQ will be used to calculate descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the LOQ).

If methods based on the assumption that the data are normally distributed are not adequate, analyses may be performed on transformed data or nonparametric analysis methods may be used, as appropriate.

Natural logarithm transformation will be used for plasma/blood concentrations and analysis of PK parameters. Plasma concentration values that are below the limit of quantitation (BLQ) will be presented as "BLQ" in the concentration data listing. Values that are BLQ will be treated as 0 at predose time points, and one-half the value of the LOQ at postbaseline time points.

The following conventions will be used for the presentation of summary and order statistics:

- If at least 1 subject has a concentration value of BLQ for the time point, the minimum value will be displayed as "BLQ."
- If more than 25% of the subjects have a concentration data value of BLQ for a given time point, the minimum and Q1 values will be displayed as "BLQ."
- If more than 50% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, and median values will be displayed as "BLQ."
- If more than 75% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, median, and Q3 values will be displayed as "BLQ."
- If all subjects have concentration data values of BLQ for a given time point, all order statistics (minimum, Q1, median, Q3, and maximum) will be displayed as "BLQ."

PK parameters that are BLQ will be imputed as one-half LOQ before log transformation or statistical model fitting.

#### 3.8. Analysis Visit Windows

#### 3.8.1. Definition of Study Day

Study day will be calculated from the first dosing date of study drug and derived as follows:

- For postdose study days: Assessment Date First Dosing Date + 1
- For days prior to the first dose: Assessment Date First Dosing Date

Therefore, study day 1 is the day of the first dose of study drug administration.

## 3.8.2. Analysis Visit Windows

The nominal visit as recorded on the CRF will be used when data are summarized by visit. Any data relating to unscheduled visits will not be assigned to a particular visit or time point. However, the following exceptions will be made:

- An unscheduled visit prior to the first dosing of study drug may be included in the calculation of the baseline value, if applicable.
- Unscheduled visits after the first dose of study drug will be included in determining the maximum postbaseline toxicity grade.
- For subjects who prematurely discontinue from the study, early termination (ET) data will be
  assigned to what would have been the next scheduled visit where the respective data were
  scheduled to be collected.
- Data collected on a follow-up visit will be summarized as a separate visit, and labeled "Follow-up Visit."
- Data obtained after the follow-up visit or last dose date plus 30 days (whichever is later) will be excluded from the summaries, but will be included in the listings.

# 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require 1 value per analysis window.

If multiple valid, nonmissing, continuous measurements exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

- In general, the baseline value will be the last nonmissing value on or prior to the first dosing date of study drug, unless specified differently. If multiple measurements occur on the same day, the last nonmissing value prior to the time of first dosing of study drug will be considered as the baseline value. If these multiple measurements occur at the same time or the time is not available, the last measurements (for continuous data) will be considered the baseline value.
- For postbaseline values:
  - The record closest to the nominal day for that visit will be selected.
  - If there are 2 records that are equidistant from the nominal day, the later record will be selected.
  - If there is more than 1 record on the selected day, the average will be taken, unless otherwise specified.

#### 4. SUBJECT DISPOSITION

#### 4.1. Subject Enrollment and Disposition

A summary of subject disposition will be provided by study group and dose level. This summary will present the number of subjects screened, the number of subjects enrolled, and the number of subjects in each of the categories listed below for each study group:

- Full Analysis Set
- Discontinued study drug with reasons for premature discontinuation of study drug
- Completed study
- Discontinued the study with reasons for premature discontinuation of study

For the status of study drug and study completion and reasons for premature discontinuation, the number and percentage of subjects in each category will be provided. The denominator for the percentage calculation will be the total number of subjects in the FAS corresponding to that column.

The following by-subject listing will be provided by subject identification (ID) number in ascending order to support the above summary tables:

• Reasons for premature study drug or study discontinuation

#### 4.2. Extent of Study Drug Exposure and Adherence

Extent of exposure to GS-5829 will be examined by assessing the total duration of exposure to study drug and the level of adherence to the study drug specified in the protocol.

## 4.2.1. **Duration of Exposure to Study Drug**

Total duration of exposure to GS-5829 will be defined as last dosing date minus first dosing date plus 1, regardless of any temporary interruptions in study drug administration, and will be expressed in weeks using up to 1 decimal place (eg, 4.5 weeks).

If the last study drug dosing date is missing,

- If the study drug is permanently withdrawn, the latest date among the study drug end date, clinical visit date, laboratory sample collection date, and vital signs assessment date that occurred during the on-treatment period will be used.
- If the study drug completion status is unknown, the earlier of the date of death or data cutoff date for analysis will be used.

The total duration of exposure to GS-5829 will be summarized using descriptive statistics and using the number (ie, cumulative counts) and percentage of subjects exposed through the following time periods: 1 day, 4 weeks, 8 weeks, 16 weeks, 24 weeks, 36 weeks, 48 weeks, and 60 weeks. Summaries will be provided by study group and dose level for the FAS.

No formal statistical testing is planned.

#### **4.2.2. Adherence to GS-5829**

The total number of tablets administered will be summarized using descriptive statistics.

The presumed total number of tablets administered to a subject will be determined by the data collected on the drug accountability CRF using the following formula:

Total Number of Doses Administered =

$$\left(\sum \text{No. of Doses Dispensed}\right) - \left(\sum \text{No. of Doses Returned}\right)$$

#### 4.2.2.1. On-Treatment Adherence

The level of on-treatment adherence to GS-5829 will be determined by the total amount of study drug administered relative to the total amount of study drug expected to be administered during a subject's actual on-treatment period based on the study drug regimen. Investigator-prescribed interruption, reductions and escalations as specified in the protocol will be taken into account.

The level of on-treatment adherence will be expressed as a percentage using the following formula:

On-Treatment Adherence (%) = 
$$\left(\frac{\text{Total Amount of Study Drug Administered}}{\text{Study Drug Expected to be Administered on Treatment}}\right) \times 100$$

Descriptive statistics for the level of on-treatment adherence with the number and percentage of subjects belonging to adherence categories (eg, < 75%,  $\ge 75$ ) will be provided by dose level for the FAS.

A by-subject listing of study drug administration and drug accountability will be provided separately by subject ID number (in ascending order) and visit (in chronological order).

No formal statistical testing is planned.

#### 4.3. Protocol Deviations

Protocol deviations occurring after subjects entered the study are documented during routine monitoring. The number and percentage of subjects with important protocol deviations by deviation reason (eg, nonadherence to study drug, violation of select inclusion/exclusion criteria) will be summarized by study group and dose level for the All Enrolled Analysis Set. A by-subject listing will be provided for those subjects with important protocol deviation.

## 5. BASELINE CHARACTERISTICS

## 5.1. Demographics

Subject demographic variables (ie, age, sex, race, and ethnicity) will be summarized by dose level, overall and study group using descriptive statistics for age, and using number and percentage of subjects for sex, race, and ethnicity. The summary of demographic data will be provided for the FAS.

A by-subject demographic listing, including the informed consent date, will be provided by subject ID number in ascending order.

#### 5.2. Other Baseline Characteristics

Other baseline characteristics include body weight (in kg), height (in cm), and body mass index (BMI; in kg/m²). These baseline characteristics will be summarized by dose level, overall and study group using descriptive statistics for continuous variables and using number and percentage of subjects for categorical variables. The summary of baseline characteristics will be provided for the FAS. No formal statistical testing is planned.

A by-subject listing of other baseline characteristics will be provided by subject ID number in ascending order.

#### **5.3.** Medical History

Medical history will be collected at screening for disease-specific and general conditions (ie, conditions not specific to the disease being studied).

General medical history data will not be coded, but will be listed only.

A by-subject listing of disease-specific and general medical history will be provided by subject ID number in ascending order.

#### 5.4. Prior Anticancer Therapy

Number of prior regimens and time since the completion of last regimen will be summarized by study group and dose level using descriptive statistics based on the FAS. A partial completion date will be imputed as follows:

- If day and month are missing but year is available, then the imputed day and month will be 01 Jan.
- If day is missing but the month and year are available, then the imputed day will be the first day of the month.
- Partial date will not be imputed if the year is missing.

The regimens and prior therapies that the subjects received will be summarized. The last regimen subjects received prior to study entry and the best response to the last regimen will be summarized.

Number of subjects who received prior radiation therapy will be listed.

#### 6. EFFICACY ANALYSES

## 6.1. Efficacy Endpoint

## 6.1.1. Definition of Efficacy Endpoints

## 6.1.1.1. Progression-free Survival

Progression-free survival is defined as the interval from first dosing date of study drug to the earlier of the first documentation of definitive disease progression or death from any cause. Definitive disease progression is determined based on RECIST v1.1 for solid tumors {Eisenhauer 2009} or Cheson Criteria {Cheson 2007} for lymphoma or PCWG2 for prostate cancer.

The date of definitive progression will be the time point at which progression is first identified by relevant radiographic, imaging, or clinical data. Data will be censored on the date of last adequate tumor assessment for subjects:

- who do not have documented progression or die, or
- who start new anticancer therapy before documented progression, or
- who start new anticancer therapy before death without documented progression, or
- who have  $\geq 2$  consecutive missing tumor assessments before documented progression, or
- who have  $\geq 2$  consecutive missing tumor assessments before death without documented progression

If a subject does not have a baseline tumor assessment, then PFS will be censored at Study Day 1, regardless of whether or not definitive progression or death has been observed.

When the date of initiation of anticancer therapy other than the study treatment is incomplete or missing, the following algorithm will be followed:

- If the day is missing but the month and year are available, then the imputed day will be the last day of the month.
- If day and month are missing but year is available, then the imputed day and month will be 01Jan or the last day of the month for the last adequate disease assessment if they have the same year, whichever is later.

#### 6.1.1.2. Overall Response Rate

Overall response rate is defined as the proportion of subjects who achieve best overall response (BOR) of complete response (CR) or partial response (PR) during study. The response definition of each response category is based on RECIST v1.1 for solid tumors, and Cheson Criteria for lymphoma. Subjects, who do not have sufficient baseline or on-study tumor status information to be adequately assessed for response status (ie, those with best overall response of not evaluable [NE]) or received anticancer therapy other than the study treatment prior to achieving CR or PR, will be considered as nonresponders and will be included in the denominators in calculations of response rates.

# 6.1.2. Analysis Methods for Efficacy Endpoints

## 6.1.2.1. Progression-free Survival

Progression-free survival based on investigators' assessments will be summarized using descriptive statistics by study group and dose level.

## 6.1.2.2. Overall Response Rate

Overall response rate based on investigators' assessments will be calculated along with its 95% CIs based on exact method. In the analyses of ORR, the BOR will be summarized by study group, dose level, and each response category as CR, PR, SD, PD, and NE.

#### 7. SAFETY ANALYSES

#### 7.1. Adverse Events and Deaths

## 7.1.1. Adverse Event Dictionary

Clinical and laboratory AEs will be coded using the current version of MedDRA. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset.

#### 7.1.2. Adverse Event Severity

Adverse events are graded by the investigator as Grade 1, 2, 3, 4, or 5 according to CTCAE Version 4.03. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings. The missing category will be listed last in summary presentation.

## 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE CRF to the question of "Related to Study Treatment." Relatedness will always default to the investigator's choice, not that of the medical monitor. Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show the relationship as missing.

#### 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if the AEs met the definitions of SAEs that were specified in the study protocol. SAEs captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Drug Safety and Public Health Department before data finalization.

#### 7.1.5. Treatment-Emergent Adverse Events

#### 7.1.5.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug
- Any AEs leading to premature discontinuation of study drug.

#### 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dosing date of study drug, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent. The event is considered treatment emergent if both of the following 2 criteria are met:

- The AE onset is the same as or after the month and year (or year) of the first dosing date of study drug, and
- The AE onset date is the same as or before the month and year (or year) of the date corresponding to 30 days after the date of the last dose of study drug

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dosing date of study drug, will be considered to be treatment emergent. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of study drug will be considered treatment emergent.

If the onset of the AE is incomplete and needs to be imputed, the following algorithm will be followed:

- If the day is missing but the month and year are available, then the imputed day will be the first day of the month or the first dosing date if they have the same month and year, whichever is later.
- If the day and month are missing but year is available, then the imputed day and month will be 01Jan or the first dosing date if they have the same year, whichever is later.

#### 7.1.6. Summaries of Adverse Events and Deaths

Treatment-emergent AEs will be summarized based on the FAS.

#### 7.1.6.1. Summaries of AE incidence by Severity

The number and percentage of subjects who experienced at least 1 TEAE will be provided and summarized by SOC, PT, dose level, and study group. For other AEs described below, summaries will be provided by SOC, PT, maximum severity, dose level, and study group:

- TEAEs
- TEAEs of Grade 3 or higher
- TE GS-5829-related AEs
- TE GS-5829-related AEs of Grade 3 or higher

- TE SAEs
- TE GS-5829-related SAEs
- TEAEs leading to premature discontinuation of GS-5829
- TEAEs leading to death
- TEAEs leading to temporary interruption of GS-5829
- TEAEs leading to dose reduction of GS-5829

A brief, high-level summary of AEs described above will be provided by study group and dose level and by the number and percentage of subjects who experienced the above AEs.

Multiple events will be counted only once per subject in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC and HLT within each SOC (if applicable), and then by PT in descending order of total frequency within each SOC. For summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in an individual subject during the study.

In addition to the above summary tables, TEAEs, TEAEs of Grade 3 or higher, TE treatment-related AEs, and TE SAEs will be summarized by PT only in descending order of total frequency.

In addition, data listings will be provided for the following:

- All AEs, indicating whether the event is treatment emergent
- All AEs of Grade 3 or higher
- SAEs
- Deaths
- AEs leading to death
- AEs leading to premature discontinuation of GS-5829
- AEs leading to temporary interruption of GS-5829
- AEs leading to dose reduction of GS-5829

## 7.1.7. Additional Analysis of Adverse Events

## 7.1.7.1. Dose Limiting Toxicity

A listing of the DLT AEs will be provided by study group and cohort including cohort number with dose level, subject identification, DLT term from investigator as well as CTCAE term and associated severity grade, if available.

#### 7.1.7.2. Treatment-Emergent Adverse Events (TEAE) of Interest

The treatment-emergent AEs of interest (AEI) include:

- Decreased Platelets (Preferred terms are defined in Appendix 2 of this SAP)
- Haemorrhage (Preferred terms are defined in Appendix 3 of this SAP)
- Diarrhoea (Preferred terms are defined in Appendix 4 of this SAP)

The AEIs will be summarized similarly to TEAE by study group and dose level cohort.

## 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the FAS and will include data collected up to the last dose of study drug plus 30 days for subjects who have permanently discontinued study drug. The analysis will be based on values reported in conventional units. When values are below the LOQ, they will be listed as such, and the closest imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7.

A by-subject listing for laboratory test results will be provided by subject ID number and visit in chronological order for hematology, serum chemistry, coagulation, and urinalysis separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on the CTCAE severity grade will be flagged in the data listings, as appropriate.

No formal statistical testing is planned.

#### 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics will be provided by study group and dose level for each laboratory test specified in the study protocol as follows:

- Baseline values
- Values at each postbaseline visit
- Change from baseline at each postbaseline visit

A baseline laboratory value will be defined as the last measurement obtained on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the visit value minus the baseline value. The mean, median, Q1, Q3, minimum, and maximum values will be displayed to the reported number of digits; StD values will be displayed to the reported number of digits plus 1.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

## 7.2.2. Graded Laboratory Values

The CTCAE, Version 4.03, will be used to assign toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (ie, increased, decreased) will be presented separately. Local labs will be graded based on central lab normal ranges with in-house macro. In the event that both central and local lab results are collected in the clinical database, the worst toxicity grade will be used for the summary of lab toxicities. All central and local laboratory values will be listed.

## 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days for subjects who permanently discontinued study drug, or the last available date in the database snapshot for subjects who were still on treatment at the time of an interim analysis. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent.

#### 7.2.2.2. Summaries of Laboratory Abnormalities

Laboratory data that are categorical will be summarized using the number and percentage of subjects in the study with the given response at baseline and each scheduled postbaseline visit.

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by lab test, dose level, and study group; subjects will be categorized according to the most severe postbaseline abnormality grade for a given lab test:

#### • Graded laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects in the FAS.

A by-subject listing of treatment-emergent laboratory abnormalities will be provided by subject ID number and visit in chronological order. This listing will include all test results that were collected throughout the study for the lab test of interest, with all applicable severity grades displayed.

## 7.2.3. Liver-related Laboratory Evaluations

Liver-related abnormalities after initial study drug dosing will be examined and summarized using the number and percentage of subjects who were reported to have the following laboratory test values for postbaseline measurements:

- Aspartate aminotransferase (AST): (a) > 3 times of the upper limit of reference range (ULN); (b) > 5 x ULN; (c) > 10 x ULN; (d) > 20 x ULN
- Alanine aminotransferase (ALT): (a) > 3 x ULN; (b) > 5 x ULN; (c) > 10 x ULN; (d) > 20 x ULN
- AST or ALT: (a)  $> 3 \times ULN$ ; (b)  $> 5 \times ULN$ ; (c)  $> 10 \times ULN$ ; (d)  $> 20 \times ULN$
- Total bilirubin: (a)  $> 1 \times ULN$ ; (b)  $> 2 \times ULN$
- Alkaline phosphatase (ALP) > 1.5 x ULN
- AST or ALT > 3 x ULN: (a) total bilirubin > 1.5 x ULN; (b) total bilirubin > 2 x ULN;
   (c) total bilirubin > 2 x ULN and ALP < 2 x ULN</li>

The summary will include data from all postbaseline visits up to 30 days after the last dose of study drug. For individual laboratory tests, subjects will be counted once based on the most severe postbaseline values. For both the composite endpoint of AST or ALT and total bilirubin, subjects will be counted once when the criteria are met at the same postbaseline visit date. The denominator is the number of subjects in the FAS who have nonmissing postbaseline values of all relevant tests at the same postbaseline visit date.

In addition, a listing of subjects who met at least 1 of the above criteria will be provided.

#### 7.2.4. Shifts Relative to the Baseline Value

Shift tables will be presented by showing change in severity grade from baseline to the worst grade postbaseline.

## 7.3. Body Weight and Vital Signs

Descriptive statistics will be provided by study group and dose level for body weight and vital signs as follows:

- Baseline value
- Values at each postbaseline visit
- Change from baseline at each postbaseline visit

A baseline value will be defined as the last available value collected on or prior to the date of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value. Body weight and vital signs measured at unscheduled visits will be included for the baseline value selection.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3. No formal statistical testing is planned.

A by-subject listing of vital signs will be provided by subject ID number and visit in chronological order. Body weight will be included in the vital signs listing, if space permits. If not, they will be provided separately.

#### 7.4. Prior and Concomitant Medications

Medications collected at screening and during the study will be coded using the current version of the World Health Organization (WHO) Drug dictionary.

#### 7.4.1. Prior Medications

Prior medications are defined as any medications taken before a subject took the first study drug.

A summary of prior medications will not be provided.

#### 7.4.2. Concomitant Medications

Concomitant medications are defined as medications taken while a subject took study drug. Use of concomitant medications will be summarized by preferred name using the number and percentage of subjects for each study group and dose level. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered by preferred term in descending overall frequency. For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medications with a start date prior to or on the first dosing date of study drug and continued to be taken after the first dosing date, or started after the first dosing date but prior to or on the last dosing date of study drug will be considered concomitant medications. Medications started and stopped on the same day as the first dosing date or the last dosing date of study drug will also be considered concomitant. Medications with a stop date prior to the date of first dosing date of study drug or a start date after the last dosing date of study drug will be excluded from the concomitant medication summary. If a partial stop date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to the date of first study drug administration will be excluded from the concomitant medication summary. If a partial start date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) after the study drug stop date will be excluded from the concomitant medication summary. Medications with completely missing start and stop dates will be included in the concomitant medication summary, unless otherwise specified. Summaries will be based on the FAS. No formal statistical testing is planned.

All prior and concomitant medications (other than per-protocol study drugs) will be provided in a by-subject listing sorted by subject ID number and administration date in chronological order.

## 7.5. Electrocardiogram Results

Electrocardiogram (ECG) analysis results are intended to identify meaningful changes in the QT interval. If potential abnormalities of interest are identified, further analyses may be conducted. Summaries of ECG data will be provided for the FAS for each scheduled time point. Both central and local ECG measurements will be considered for analysis. No formal statistical testing is planned.

#### 7.5.1. Corrected QT Intervals

The QT interval (measured in millisecond [msec]) is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. The QT interval represents electrical depolarization and repolarization of the ventricles. The QT interval is affected by heart rate, and a number of methods have been proposed to correct QT for heart rate.

Corrected QT (QTc) intervals will be derived using Fridericia's correction (QTcF) as follows:

$$QTcF = \frac{QT}{\sqrt[3]{RR}}$$

where QT is measured in msec; RR = 60/Heart Rate (beats per min [bpm]) and RR is measured in seconds

The maximum postdose QTcF interval values obtained during the study will be summarized within the following categories:

- < 450 msec
- $> 450 \text{ msec} \le 480 \text{ msec}$
- > 480 msec < 500 msec
- > 500 msec

The maximum postdose change in QTcF interval values obtained during the study will also be summarized within the following categories:

- < 30 msec
- $> 30 \text{ msec} \le 60 \text{ msec}$
- > 60 msec

The QTcF and uncorrected QT values at each visit and time point and change from baseline at each visit and time point will be summarized for the FAS by study group and dose level using descriptive statistics.

#### 7.5.2. PR and QRS Intervals

The PR interval (measured in msec) is a measure of the time between the start of the P wave (the onset of atrial depolarization) and the beginning of the QRS complex (the onset of ventricular depolarization). The QRS interval measures the duration of the QRS complex. The maximum ventricular rate (VR) and PR and QRS intervals observed during the study will be categorized. The number and percentage of subjects having values in the following ranges will be presented by study group and dose level:

- VR > 100 bpm
- PR interval > 200 msec
- QRS interval > 110 msec

In addition, VR, PR, RR, and QRS values at each visit and time point and change from baseline at each visit and time point will be summarized for the FAS by study group and dose level using descriptive statistics.

## 7.6. Other Safety Measures

No additional safety measures are specified in the protocol.

## 7.7. Changes From Protocol-Specified Safety Analyses

There are no deviations from the protocol-specified safety analyses.

# 8. PHARMACOKINETIC (PK) ANALYSES

## 8.1. PK Sample Collection

Plasma samples for GS-5829 PK will be collected in cohorts 1 - 3 of Group 1 on Study Day 1 at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose and in cohorts 4 - 6 of Group 1 and all cohorts of Group 2 on Cycle 1 Day 1 at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose. Additional samples will be collected at 48 and 72 hours postdose in cohorts 1 - 3 of Group 1 relative to first dose of GS-5829. Plasma samples for GS-5829 PK will be collected in all cohorts at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post dose relative to GS-5829 administration on Cycle 1 Day 8. Sparse PK samples will be collected in all cohorts at trough (20 - 26 hours postdose) on Cycle 1 Day 4, 2 - 4 hours post dose on Cycle 1 Day 15, and anytime postdose on Day 1 of Cycles 2 through 6. In one or more cohorts, PK samples will be collected on Day 1 of Cycle 2 at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post dose.

#### 8.1.1. Estimation of PK Parameters

PK parameters will be estimated using Phoenix WinNonlin® software using standard noncompartmental methods. The linear/log trapezoidal rule will be used in conjunction with the appropriate noncompartmental model, with input values for dose level, dosing time, plasma concentration, and corresponding real-time values, based on drug dosing times whenever possible.

All predose sample times before time-zero will be converted to 0.

For area under the curve (AUC), samples BLQ of the bioanalytical assays occurring prior to the achievement of the first quantifiable concentration will be assigned a concentration value of 0 to prevent overestimation of the initial AUC. Samples that are BLQ at all other time points will be treated as missing data in WinNonlin. The nominal time point for a key event or dosing interval  $(\tau)$  may be used to permit direct calculation of AUC over specific time intervals. The appropriateness of this approach will be assessed by the PK scientist on a profile-by-profile basis.

Pharmacokinetic parameters such as  $AUC_{tau}$ ,  $\lambda_z$  and  $t_{1/2}$  are dependent on an accurate estimation of the terminal elimination phase of drug. The appropriateness of calculating these parameters will be evaluated upon inspection of PK data on a profile-by-profile basis by the PK scientist.

#### 8.1.2. PK Parameters

PK parameters will be generated for all subjects in the PK analysis set. The analytes presented in Table 1 will be evaluated if data are available.

| | GS-5829 | GS-697412 | Metabolite/parent ratio |
|---|---|---|---|
| Study Day 1/ Cycle 1 Day 1<br>(Study Day 1 only applies to<br>Group 1 cohort 1-3) | $C_{max}, T_{max}, AUC_{0\text{-}24h}, \\ AUC_{last}, AUC_{inf}, C_{24h}, \\ C_{last}, T_{last}, \lambda_z, T_{1/2}, \\ V_z F_obs, CL_F_obs$ | $\begin{array}{c} C_{max},T_{max},AUC_{0\text{-}24h,}\\ AUC_{last},AUC_{inf},C_{24h},C_{last},\\ T_{last},\lambda_z,T_{1/2} \end{array}$ | $C_{\text{max}}$ , $AUC_{0\text{-}24h}$ , and $C_{24h}$ |
| Cycle 1 Day 8 | $\begin{array}{c} C_{max}, T_{max}, AUC_{tau,} \\ AUC_{last}, AUC_{inf}, C_{tau}, \\ C_{last}, T_{last}, \lambda_z, T_{1/2}, V_z\_F, \\ CL_{ss}\_F \end{array}$ | $\begin{array}{c} C_{max}, T_{max}, AUC_{tau,}\\ AUC_{last}, AUC_{inf}, C_{tau}, C_{last},\\ T_{last}, \lambda_z, T_{1/2} \end{array}$ | $C_{max}$ , $AUC_{tau}$ , and $C_{tau}$ |

**Table 1.** PK Parameters for Analytes

Individual subject concentration data and individual subject PK parameters for GS-5829 and its metabolite GS-697412 will be listed and summarized using descriptive statistics by treatment. Summary statistics (n, mean, StD, coefficient of variation [%CV], median, min, max, Q1, and Q3) will be presented for both individual subject concentration data by time point and individual subject PK parameters by dose level. Moreover, the geometric mean, 95% CI, and the mean and StD of the natural log-transformed values will be presented for individual subject PK parameter data.

Individual metabolite to parent ratios will be calculated for  $AUC_{0-24h}$ ,  $C_{max}$ , and  $C_{24h}$  on Study Day 1 and Cycle 1 Day 1, and for  $AUC_{tau}$ ,  $C_{max}$ , and  $C_{tau}$  on Cycle 1 Day 8, when available, and summarized similarly to the PK parameters.

Individual concentration data listings and summaries will include all subjects with concentration data. The sample size for each time point will be based on the number of subjects with nonmissing concentration data at that time point. The number of subjects with concentration BLQ will be presented for each time point. For summary statistics, BLQ values will be treated as 0 at predose and one-half of the lower limit of quantitation (LLOQ) for postdose time points.

Individual PK parameter data listings and summaries will include all subjects for whom PK parameter(s) can be derived. The sample size for each PK parameter will be based on the number of subjects with nonmissing data for that PK parameter.

The following tables will be provided by dose level:

- Individual subject concentration data and summary statistics
- Individual subject plasma PK parameters and summary statistics
- Individual metabolite to parent ratios for  $AUC_{0-24h}$ ,  $C_{max}$ , and  $C_{24h}$  on Study Day 1 and Cycle 1 Day 1, and for  $AUC_{tau}$ ,  $C_{max}$ , and  $C_{tau}$ , on Cycle 1 Day 8 and its summary statistics.

The following figures may be provided by dose level:

- Mean (± StD) concentration data versus time (on linear and semilogarithmic scales)
- Median (Q1, Q3) concentration data versus time (on linear and semilogarithmic scales)

Individual, mean, and median postdose concentration values that are  $\leq$  LLOQ will not be displayed in the figures and remaining points connected.

PK sampling details by subject, including procedures, differences in scheduled and actual draw times, and sample age will be provided in listings.

# 9. REFERENCES

- Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, et al. Revised response criteria for malignant lymphoma. J Clin Oncol 2007;25 (5):579-86.
- Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New Response Evaluation Criteria in Solid Tumours: Revised RECIST Guideline (Version 1.1). Eur J Cancer 2009;45 (2):228-47.
- Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, et al. Design and End Points of Clinical Trials for Patients With Progressive Prostate Cancer and Castrate Levels of Testosterone: Recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol 2008;26 (7):1148-59.

# 10. SOFTWARE

SAS® Software Version 9.4. SAS Institute Inc., Cary, NC, USA.

# 11. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
## 12. APPENDICES

## **Appendix 1.** Schedule of Assessments

| | | | First 28 Days | | | | | | | | Cycle 2 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Phase Cycle Day | Screening<br>Day 28 | Study<br>Day 1 <sup>a</sup> | Cycle 1<br>Day 1 <sup>b</sup> | Day 2 | Day 4 | Day 8 | Day 11 | Day 15 | Day 22 | Cycle 2 Day 1 and Every 2 weeks* | Day 1<br>and<br>Every<br>4 weeks | Every<br>8 weeks | ЕОТ | 30 day<br>Safety<br>Follow-up <sup>k</sup> |
| Window (day) | -28 | ±0 | ±3 | ±0 | ±0 | ±1 | ±1 | ±2 | ±3 | ±7 | ±7 | ±7 | ±7 | ±7 |
| Informed Consent | X | | | | | | | | | | | | | |
| Medical and Medication<br>History <sup>c</sup> | X | | | | | | | | | | | | | |
| Physical Examination <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | | | X | |
| Vital Signs <sup>e</sup> | X | X | X | X | X | X | X | X | X | X | | | X | |
| Oxygen saturation <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | | | X | |
| Echocardiogram <sup>r</sup> | X | | | | | | | | | | X | | X | |
| Triplicate 12-lead ECG <sup>g</sup> | X | X | X | | | X | | | | | X | | X | |
| Adverse events/<br>Concomitant medications <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | | | X | X |
| IP Dispensing | | $X^{i}$ | X | | | | | | | | X | | | |
| Exemestane or Fulvestrant <sup>w</sup> (Group 2 only) | | | X | | | | | X | | | X | | | |
| Dosing Diary Accountability | | | X | X | X | X | X | X | X | X | | | | |
| IXRS Registration | X | X | $X^{j}$ | | | | | | | X | | | X | |
| CBC with differential | X <sup>s</sup> | X | X | | X | X | X | X | X | X | | | X | |
| Chemistry <sup>y</sup> | X <sup>s</sup> | X | X | | X | X | X | X | X | X | | | X | |
| Coagulation <sup>q</sup> | X <sup>s</sup> | | X | | | X | | | | | X | | X | |
| 25-hydroxy vitamin D<br>(Group 2 only) | X | | | | | | | | | | | | | |

| | | | First 28 Days | | | | | | | Cycle 2 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Phase Cycle Day | Screening<br>Day 28 | Study<br>Day 1 <sup>a</sup> | Cycle 1<br>Day 1 <sup>b</sup> | Day 2 | Day 4 | Day 8 | Day 11 | Day 15 | Day 22 | Cycle 2 Day 1 and Every 2 weeks* | Day 1<br>and<br>Every<br>4 weeks | Every<br>8 weeks | ЕОТ | 30 day<br>Safety<br>Follow-up <sup>k</sup> |
| Window (day) | -28 | ±0 | ±3 | ±0 | ±0 | ±1 | ±1 | ±2 | ±3 | ±7 | ±7 | ±7 | ±7 | ±7 |
| Urinalysis and Urine<br>Chemistry | | X | X | | | X | | | X | X | | | X | |
| Pregnancy Test <sup>1</sup> | X | X | $X^{j}$ | | | | | | | | X | | X | |
| GS-5829 Intensive PK <sup>m</sup> | | X | X | | | X | | | | | X <sup>v</sup> | | | |
| GS-5829 Sparse PK <sup>m</sup> | | | | | X | | | X | | | X <sup>v</sup> | | | |
| CCI | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | ' | | | |
| CCI | | | | | | | | | | | | | | |
| Biopsies for Group 3<br>lymphoma expansion <sup>x</sup> | X | | | | | | | | | X <sup>x</sup> | | | X | |
| CT Scan w/Contrast or MRI <sup>P</sup> | X | | | | | | | | | | | X | X <sup>P</sup> | |
| PET Scan (Group 3 only) <sup>z</sup> | X | | | | | | | | | | | | | |
| Bone Scan(Group 2 only) | X | | | | | | | | | | | | X | |
| ECOG Performance Status | X | X | X | | | X | | X | X | | | | X | |
| Treatment Response<br>Assessment <sup>t</sup> | | | | | | | | | | | | X | X | |

<sup>\*</sup> Day 1 of subsequent cycles.

a Study Day 1 is applicable to Cohorts 1-3 only of Group 1.

b Cycle 1 Day 1 occurs on Study Day 7 for subjects in Cohorts 1-3 of Group 1 and must occur at least 5 days, but no more than 9 days after Study Day 1. For Group 1 Cohorts 4 and higher and all cohorts of Group 2 the first day of study is Cycle 1 Day 1.

c Medical history includes significant past medical events (eg, prior hospitalizations or surgeries), a review of the disease under study, prior anti-cancer therapies, and any concurrent medical illnesses.

d Screening and End of Treatment Physical Examinations (PE) will be a complete PE. Beginning at Study Day 1 (Group 1 Cohorts 1-3) and C1D1 (all groups), a modified physical examination will be performed to monitor for any changes (e.g. lymph nodes, lung, cardiac, abdomen, skin, neurologic, and any systems, as clinically indicated). Weight (without shoes) should be measured at each PE. Height (without shoes) should be measured at screening only.

- e Study Day 1 (Cohorts 1-3 of Group 1) and C1D1 (all groups) vital signs will be taken within 15 min pre-GS-5829 dose. C1D1 vitals will also be collected at 2 and 4 hours post dose (+/- 15 min); vital signs will be taken pre-dose only at all subsequent visits.
- f Oxygen saturation will be tested with a pulse oximeter.
- g ECG: At Screening, at predose on Day 1 of each Cycle starting with Cycle 2, and at EOT, a triplicate 12-lead ECG will be collected at a single timepoint. On Study Day 1(Cohorts 1-3 only) and C1D1 (Cohorts 4-8 only and all cohorts of Group 2), C1D8 (all cohorts) (at predose, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, and 12 hours post first dose +/- 20 min) and Day 1 of cycles 2-6 (at pre-dose). Subjects in the Group 3 lymphoma expansion will have ECGs collected at pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Cycle 1, Day 8. ECGs will also be collected at pre-dose on Day 1 of Cycles 2, 4, and 6. ECGs should always be collected prior to PK (or any other blood draw) if they are to be collected at the same nominal timepoint. Subjects should be resting quietly and free of distraction (eg, TV, conversation) for 10 minutes prior to ECG collection and ECGs should be collected over a 5 minute window at each timepoint.
- h Adverse events will be assessed at pre- and post-GS-5829 dosing during applicable clinic visits. Subjects will also return to clinic at 30-day post last IP dose, to assess AEs and SAEs.
- i Cohorts 1-3 of Group 1 will receive one dose of GS-5829 on Study Day 1, which will be administered in the clinic.
- j Not applicable to subjects in Cohort 1-3 of Group 1.
- k Subjects who miss the 30 day Safety Follow-up visit will be contacted by phone 30 days (± 2 days) after the last dose of GS-5829 to assess AEs.
- 1 If applicable (females of child bearing potential). Serum pregnancy will be conducted at Screening. Urine pregnancy will be conducted pre-dose on Study Day 1/C1D1 of each cycle and at EOT.
- m Plasma samples for GS-5829 PK will be collected (± 10 minutes) in cohorts 1-3 of Group 1 on Study Day 1 at pre-dose (0 hr), 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose, and in cohorts 4-8 of Group 1 and all cohorts of Group 2 on Cycle 1 Day 1 at pre-dose (0 hr), 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose. Additional samples will be collected at 48 and 72 hours post-dose in cohorts 1 3 of Group 1 relative to first dose of GS-5829. Plasma samples for GS-5829 PK will be collected in all cohorts (Group 1 and Group 2) at pre-dose (0 hr), 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose relative to GS-5829 administration on Cycle 1 Day 8. Sparse PK samples will be collected in all cohorts (Group 1 and Group 2) at trough (20-26 hours post-dose) on Cycle 1 Day 4, 2 4 hours post-dose on Cycle 1 Day 15, and anytime post-dose on Day 1 of Cycles 2 through 6. Urine will be collected for GS-5829 PK in Group 1 cohorts 1-3 on Study Day 1 and in Group 1 cohorts 4-8 on Cycle 1 Day 1 at pre-dose (0 hr), 0-6 hours, 6-12 hours, and 12-24 hours post-dose relative to first dose of GS-5829. Subjects in the Group 3 lymphoma expansion will have PK drawn at pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Cycle 1, Day 8. PK samples will also be drawn at pre-dose on Day 1 of Cycles 2, 4, and 6

- Tumor evaluation by CT/MRI or applicable scan will be performed during screening (within 28 days of Day 1) and every 8 weeks thereafter for the first year and then every 12 weeks. A baseline scan within 8 weeks of Day 1 is acceptable. The same radiographic procedure used to define measurable lesions must be used throughout the study for each subject. CT/MRI or applicable scan should be conducted at the EOS visit if not conducted within the previous 4 weeks. Subjects with prostate cancer or in Group 2 should also undergo a bone scan. Scan at EOT visit is not necessary if restaging scan is performed within 4 weeks of the EOT.
- q Includes PT/PTT.
- Echocardiogram will be performed at screening, C2D1, and EOT. MUGA is acceptable. The same modality must be used throughout study participation.
- s Screening chemistry, hematology and coagulation to be collected within 7 days of Study Day 1/C1D1.
- t Bone marrow biopsy is only to be performed to assess suspected CR, and only if the subject had lymphoma involvement of the marrow at baseline (or did not have a baseline marrow biopsy). After CR is determined, there is no need for any further bone marrow biopsy assessments.
- At one or more dose levels, GS-5829 will be administered in fed state on Day 1 of Cycle 2 and PK samples will be collected at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose. In subjects where intensive PK is collected on Cycle 2, Day 1, sparse PK samples do not need to be collected at that visit.

- w Subjects assigned to receive exemestane in combination with GS-5829 in the study will self-administer exemestane orally once daily starting on or before on Cycle 1 Day 1 and thereafter at approximately the same time each day until the end of treatment. Subjects assigned to receive fulvestrant in combination with GS-5829 in this study will receive fulvestrant 500 mg IM on Cycle 1 Day 1 and every 28 days (+/- 3 days) until the end of treatment. For subjects initiating fulvestrant on this study a single dose of fulvestrant 500 mg should be administered on Cycle 1 Day 15 (+/- 3 days).
- x Biopsies are requested from subjects with accessible disease and should be core needle or excision biopsies. The pre-treatment biopsy can be obtained any time after the last line of therapy and prior to the first dose, the Cycle 2 Day 15 biopsy can be obtained anytime between Cycle 2 Day 1 and Cycle 2Day 21. The EOT biopsy should be collected at progression only for subjects with progressive disease.
- y AAG will be collected at Screening, pre-dose on C1D1 and C1D8 only. Ferritin and CRP will be collected pre-dose on C1D1 and Day 1 of every subsequent cycle.
- z Subjects who are enrolled in Group 3 will undergo a baseline PET/CT scan and at Week 16 in the place of a CT scan if available.

**Appendix 2.** List of Medical Search Terms for Decreased Platelets

| MEDDRA Term Name | MEDDRA Code |
|----------------------------------------------------|-------------|
| Amegakaryocytic thrombocytopenia | 10076744 |
| Cutaneovisceral angiomatosis with thrombocytopenia | 10069098 |
| HELLP syndrome | 10049058 |
| Immune thrombocytopenic purpura | 10074667 |
| Platelet production decreased | 10035540 |
| Thrombocytopenia | 10043554 |
| Thrombocytopenic purpura | 10043561 |
| Thrombotic thrombocytopenic purpura | 10043648 |
| Severe fever with thrombocytopenia syndrome | 10078387 |
| Acquired amegakaryocytic thrombocytopenia | 10076747 |
| Megakaryocytes decreased | 10027119 |
| Platelet count decreased | 10035528 |
| Platelet maturation arrest | 10035537 |
| Platelet production decreased | 10035540 |
| Platelet toxicity | 10059440 |
| Thrombocytopenia | 10043554 |
| Megakaryocytes abnormal | 10027118 |
| Platelet count abnormal | 10035526 |
| Platelet disorder | 10035532 |
| Plateletcrit abnormal | 10064785 |
| Plateletcrit decreased | 10064784 |
| Thrombocytopenia neonatal | 10043557 |

**Appendix 3.** List of Medical Search Terms for Haemorrhage

| MEDDRA Term Name | MEDDRA Code |
|---|---|
| Haemorrhagic adrenal infarction | 10079902 |
| Eye haematoma | 10079891 |
| Spontaneous hyphaema | 10080110 |
| Anal fissure haemorrhage | 10079765 |
| Paranasal sinus haemorrhage | 10080108 |
| Peripheral artery aneurysm rupture | 10079908 |
| Aortic annulus rupture | 10079586 |
| Abdominal wall haematoma | 10067383 |
| Abdominal wall haemorrhage | 10067788 |
| Abnormal clotting factor | 10049862 |
| Abnormal withdrawal bleeding | 10069195 |
| Acquired dysfibrinogenaemia | 10051122 |
| Acquired haemophilia | 10053745 |
| Acquired haemophilia with anti FVIII, XI, or XIII | 10056496 |
| Acquired protein S deficiency | 10068370 |
| Acquired Von Willebrand's disease | 10069495 |
| Activated partial thromboplastin time abnormal | 10000631 |
| Activated partial thromboplastin time prolonged | 10000636 |
| Activated partial thromboplastin time ratio abnormal | 10075284 |
| Activated partial thromboplastin time ratio fluctuation | 10075286 |
| Activated partial thromboplastin time ratio increased | 10075287 |
| Acute haemorrhagic leukoencephalitis | 10058994 |
| Acute haemorrhagic ulcerative colitis | 10075634 |
| Administration site bruise | 10075094 |
| Administration site haematoma | 10075100 |
| Administration site haemorrhage | 10075101 |
| Adrenal haematoma | 10059194 |
| Adrenal haemorrhage | 10001361 |
| Anal haemorrhage | 10049555 |
| Anal ulcer haemorrhage | 10063896 |
| Anastomotic haemorrhage | 10056346 |

| MEDDRA Term Name | MEDDRA Code |
|----------------------------------------|-------------|
| Anastomotic ulcer haemorrhage | 10002244 |
| Aneurysm ruptured | 10048380 |
| Angina bullosa haemorrhagica | 10064223 |
| Anorectal varices haemorrhage | 10068925 |
| Anti factor IX antibody positive | 10058748 |
| Anti factor V antibody positive | 10058745 |
| Anti factor VII antibody positive | 10058746 |
| Anti factor VIII antibody positive | 10049013 |
| Anti factor X activity abnormal | 10077670 |
| Anti factor X activity increased | 10077671 |
| Anti factor X antibody positive | 10058747 |
| Anti factor XI antibody positive | 10058749 |
| Anti factor XII antibody positive | 10058750 |
| Antithrombin III increased | 10051115 |
| Aortic aneurysm rupture | 10002886 |
| Aortic dissection rupture | 10068119 |
| Aortic intramural haematoma | 10067975 |
| Aortic perforation | 10075729 |
| Aortic rupture | 10060874 |
| Aponeurosis contusion | 10075330 |
| Application site bruise | 10050114 |
| Application site haematoma | 10068317 |
| Application site haemorrhage | 10072694 |
| Application site purpura | 10050182 |
| Arterial haemorrhage | 10060964 |
| Arterial intramural haematoma | 10074971 |
| Arterial ligation | 10003165 |
| Arterial perforation | 10075732 |
| Arterial rupture | 10003173 |
| Arteriovenous fistula site haematoma | 10055150 |
| Arteriovenous fistula site haemorrhage | 10055123 |
| Arteriovenous graft site haematoma | 10055152 |

| MEDDRA Term Name | MEDDRA Code |
|--------------------------------------|-------------|
| Arteriovenous graft site haemorrhage | 10055126 |
| Atrial rupture | 10048761 |
| Auricular haematoma | 10003797 |
| Basal ganglia haematoma | 10077031 |
| Basal ganglia haemorrhage | 10067057 |
| Basilar artery perforation | 10075736 |
| Benign familial haematuria | 10060876 |
| Bladder tamponade | 10062656 |
| Bleeding time abnormal | 10049227 |
| Bleeding time prolonged | 10005140 |
| Bleeding varicose vein | 10005144 |
| Blood blister | 10005372 |
| Blood fibrinogen abnormal | 10005518 |
| Blood fibrinogen decreased | 10005520 |
| Blood thrombin abnormal | 10005818 |
| Blood thrombin decreased | 10005820 |
| Blood thromboplastin abnormal | 10005824 |
| Blood thromboplastin decreased | 10005826 |
| Blood urine | 10005863 |
| Blood urine present | 10018870 |
| Bloody discharge | 10057687 |
| Bloody peritoneal effluent | 10067442 |
| Bone contusion | 10066251 |
| Bone marrow haemorrhage | 10073581 |
| Brain contusion | 10052346 |
| Brain stem haematoma | 10073230 |
| Brain stem haemorrhage | 10006145 |
| Brain stem microhaemorrhage | 10071205 |
| Breast haematoma | 10064753 |
| Breast haemorrhage | 10006254 |
| Broad ligament haematoma | 10006375 |
| Bronchial haemorrhage | 10065739 |

| MEDDRA Term Name | MEDDRA Code |
|--------------------------------------------------|-------------|
| Bronchial varices haemorrhage | 10079163 |
| Bursal haematoma | 10077818 |
| Capillary fragility abnormal | 10007192 |
| Capillary fragility increased | 10007194 |
| Capillary permeability increased | 10007200 |
| Cardiac contusion | 10073356 |
| Carotid aneurysm rupture | 10051328 |
| Carotid artery perforation | 10075728 |
| Catheter site bruise | 10063587 |
| Catheter site haematoma | 10055662 |
| Catheter site haemorrhage | 10051099 |
| Central nervous system haemorrhage | 10072043 |
| Cephalhaematoma | 10008014 |
| Cerebellar haematoma | 10061038 |
| Cerebellar haemorrhage | 10008030 |
| Cerebellar microhaemorrhage | 10071206 |
| Cerebral aneurysm perforation | 10075394 |
| Cerebral aneurysm ruptured syphilitic | 10008076 |
| Cerebral arteriovenous malformation haemorrhagic | 10008086 |
| Cerebral artery perforation | 10075734 |
| Cerebral haematoma | 10053942 |
| Cerebral haemorrhage | 10008111 |
| Cerebral haemorrhage foetal | 10050157 |
| Cerebral haemorrhage neonatal | 10008112 |
| Cerebral microhaemorrhage | 10067277 |
| Cervix haematoma uterine | 10050020 |
| Cervix haemorrhage uterine | 10050022 |
| Chest wall haematoma | 10076597 |
| Choroidal haematoma | 10068642 |
| Choroidal haemorrhage | 10008786 |
| Chronic gastrointestinal bleeding | 10050399 |
| Chronic pigmented purpura | 10072726 |

| MEDDRA Term Name | MEDDRA Code |
|-----------------------------------------|-------------|
| Ciliary body haemorrhage | 10057417 |
| Circulating anticoagulant | 10053627 |
| Clot retraction abnormal | 10009669 |
| Clot retraction time prolonged | 10009675 |
| Coagulation disorder neonatal | 10009732 |
| Coagulation factor decreased | 10009736 |
| Coagulation factor deficiency | 10067787 |
| Coagulation factor IX level abnormal | 10061770 |
| Coagulation factor IX level decreased | 10009746 |
| Coagulation factor mutation | 10065442 |
| Coagulation factor V level abnormal | 10061771 |
| Coagulation factor V level decreased | 10009754 |
| Coagulation factor VII level abnormal | 10061772 |
| Coagulation factor VII level decreased | 10009761 |
| Coagulation factor VIII level abnormal | 10061773 |
| Coagulation factor VIII level decreased | 10009768 |
| Coagulation factor X level abnormal | 10061774 |
| Coagulation factor X level decreased | 10009775 |
| Coagulation factor XI level abnormal | 10061775 |
| Coagulation factor XI level decreased | 10009779 |
| Coagulation factor XII level abnormal | 10061776 |
| Coagulation factor XII level decreased | 10009783 |
| Coagulation factor XIII level abnormal | 10061777 |
| Coagulation factor XIII level decreased | 10009787 |
| Coagulation time abnormal | 10009791 |
| Coagulation time prolonged | 10009799 |
| Coagulopathy | 10009802 |
| Coital bleeding | 10065019 |
| Colonic haematoma | 10009996 |
| Congenital coagulopathy | 10063563 |
| Congenital dysfibrinogenaemia | 10051123 |
| Conjunctival haemorrhage | 10010719 |

| MEDDRA Term Name | MEDDRA Code |
|----------------------------------------|-------------|
| Contusion | 10050584 |
| Corneal bleeding | 10051558 |
| Cullen's sign | 10059029 |
| Cystitis haemorrhagic | 10011793 |
| Deep dissecting haematoma | 10074718 |
| Diarrhoea haemorrhagic | 10012741 |
| Dilutional coagulopathy | 10060906 |
| Disseminated intravascular coagulation | 10013442 |
| Diverticulitis intestinal haemorrhagic | 10013541 |
| Diverticulum intestinal haemorrhagic | 10013560 |
| Duodenal ulcer haemorrhage | 10013839 |
| Duodenitis haemorrhagic | 10013865 |
| Dysfunctional uterine bleeding | 10013908 |
| Ear haemorrhage | 10014009 |
| Ecchymosis | 10014080 |
| Encephalitis haemorrhagic | 10014589 |
| Endometriosis | 10014778 |
| Enterocolitis haemorrhagic | 10014896 |
| Epidural haemorrhage | 10073681 |
| Epistaxis | 10015090 |
| Ethanol gelation test positive | 10062650 |
| Exsanguination | 10015719 |
| Extra-axial haemorrhage | 10078254 |
| Extradural haematoma | 10015769 |
| Extravasation blood | 10015867 |
| Eye contusion | 10073354 |
| Eye haemorrhage | 10015926 |
| Eyelid bleeding | 10053196 |
| Eyelid contusion | 10075018 |
| Eyelid haematoma | 10064976 |
| Factor I deficiency | 10016075 |
| Factor II deficiency | 10016076 |

| MEDDRA Term Name | MEDDRA Code |
|----------------------------------------|-------------|
| Factor III deficiency | 10052473 |
| Factor IX deficiency | 10016077 |
| Factor V deficiency | 10048930 |
| Factor VII deficiency | 10016079 |
| Factor VIII deficiency | 10016080 |
| Factor X deficiency | 10052474 |
| Factor Xa activity abnormal | 10078667 |
| Factor Xa activity decreased | 10078676 |
| Factor XI deficiency | 10016082 |
| Factor XII deficiency | 10051806 |
| Factor XIII deficiency | 10016083 |
| Femoral artery perforation | 10075739 |
| Femoral vein perforation | 10075745 |
| Fibrin abnormal | 10016575 |
| Fibrin D dimer decreased | 10016579 |
| Fibrin D dimer increased | 10016581 |
| Fibrin decreased | 10016584 |
| Fibrin degradation products | 10016585 |
| Fibrin degradation products increased | 10016588 |
| Fibrinolysis abnormal | 10016604 |
| Fibrinolysis increased | 10016607 |
| Foetal-maternal haemorrhage | 10016871 |
| Gardner-Diamond syndrome | 10078888 |
| Gastric haemorrhage | 10017788 |
| Gastric occult blood positive | 10067855 |
| Gastric ulcer haemorrhage | 10017826 |
| Gastric ulcer haemorrhage, obstructive | 10017829 |
| Gastric varices haemorrhage | 10057572 |
| Gastritis alcoholic haemorrhagic | 10017857 |
| Gastritis haemorrhagic | 10017866 |
| Gastroduodenal haemorrhage | 10053768 |
| Gastroduodenitis haemorrhagic | 10048712 |

| MEDDRA Term Name | MEDDRA Code |
|----------------------------------------------|-------------|
| Gastrointestinal angiectasia | 10078142 |
| Gastrointestinal angiodysplasia haemorrhagic | 10017929 |
| Gastrointestinal haemorrhage | 10017955 |
| Gastrointestinal organ contusion | 10078655 |
| Gastrointestinal polyp haemorrhage | 10074437 |
| Gastrointestinal ulcer haemorrhage | 10056743 |
| Genital contusion | 10073355 |
| Genital haemorrhage | 10061178 |
| Gingival bleeding | 10018276 |
| Graft haemorrhage | 10063577 |
| Grey Turner's sign | 10075426 |
| Haemarthrosis | 10018829 |
| Haematemesis | 10018830 |
| Haematochezia | 10018836 |
| Haematocoele | 10018833 |
| Haematoma | 10018852 |
| Haematoma evacuation | 10060733 |
| Haematoma infection | 10051564 |
| Haematosalpinx | 10050468 |
| Haematospermia | 10018866 |
| Haematotympanum | 10063013 |
| Haematuria | 10018867 |
| Haematuria traumatic | 10018871 |
| Haemobilia | 10058947 |
| Haemophilia | 10061992 |
| Haemophilia A with anti factor VIII | 10056492 |
| Haemophilia A without inhibitors | 10056493 |
| Haemophilia B with anti factor IX | 10056494 |
| Haemophilia B without inhibitors | 10056495 |
| Haemophilic arthropathy | 10065057 |
| Haemophilic pseudotumour | 10073770 |
| Haemoptysis | 10018964 |

| MEDDRA Term Name | MEDDRA Code |
|-----------------------------------------|-------------|
| Haemorrhage | 10055798 |
| Haemorrhage coronary artery | 10055803 |
| Haemorrhage foetal | 10061191 |
| Haemorrhage in pregnancy | 10018981 |
| Haemorrhage intracranial | 10018985 |
| Haemorrhage neonatal | 10061993 |
| Haemorrhage subcutaneous | 10018999 |
| Haemorrhage subepidermal | 10019001 |
| Haemorrhage urinary tract | 10055847 |
| Haemorrhagic anaemia | 10052293 |
| Haemorrhagic arteriovenous malformation | 10064595 |
| Haemorrhagic ascites | 10059766 |
| Haemorrhagic breast cyst | 10077443 |
| Haemorrhagic cerebral infarction | 10019005 |
| Haemorrhagic cyst | 10059189 |
| Haemorrhagic diathesis | 10062713 |
| Haemorrhagic disease of newborn | 10019008 |
| Haemorrhagic disorder | 10019009 |
| Haemorrhagic erosive gastritis | 10067786 |
| Haemorrhagic hepatic cyst | 10067796 |
| Haemorrhagic infarction | 10019013 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Haemorrhagic ovarian cyst | 10060781 |
| Haemorrhagic pneumonia | 10077933 |
| Haemorrhagic stroke | 10019016 |
| Haemorrhagic thyroid cyst | 10072256 |
| Haemorrhagic transformation stroke | 10055677 |
| Haemorrhagic tumour necrosis | 10054096 |
| Haemorrhagic urticaria | 10059499 |
| Haemorrhagic varicella syndrome | 10078873 |
| Haemorrhagic vasculitis | 10071252 |
| Haemorrhoidal haemorrhage | 10054787 |

| MEDDRA Term Name | MEDDRA Code |
|----------------------------------------|-------------|
| Haemostasis | 10067439 |
| Haemothorax | 10019027 |
| Henoch-Schonlein purpura | 10019617 |
| Hepatic haemangioma rupture | 10054885 |
| Hepatic haematoma | 10019676 |
| Hepatic haemorrhage | 10019677 |
| Hereditary haemorrhagic telangiectasia | 10019883 |
| Hermansky-Pudlak syndrome | 10071775 |
| Hyperfibrinolysis | 10074737 |
| Hyphaema | 10020923 |
| Hypocoagulable state | 10020973 |
| Hypofibrinogenaemia | 10051125 |
| Hypoprothrombinaemia | 10021085 |
| Hypothrombinaemia | 10058517 |
| Hypothromboplastinaemia | 10058518 |
| Iliac artery perforation | 10075731 |
| Iliac artery rupture | 10072789 |
| Iliac vein perforation | 10075744 |
| Immune thrombocytopenic purpura | 10074667 |
| Implant site bruising | 10063850 |
| Implant site haematoma | 10063780 |
| Implant site haemorrhage | 10053995 |
| Incision site haematoma | 10059241 |
| Incision site haemorrhage | 10051100 |
| Increased tendency to bruise | 10021688 |
| Induced abortion haemorrhage | 10052844 |
| Inferior vena cava perforation | 10075742 |
| Infusion site bruising | 10059203 |
| Infusion site haematoma | 10065463 |
| Infusion site haemorrhage | 10065464 |
| Injection site bruising | 10022052 |
| Injection site haematoma | 10022066 |

| MEDDRA Term Name | MEDDRA Code |
|------------------------------------------|-------------|
| Injection site haemorrhage | 10022067 |
| Instillation site bruise | 10073630 |
| Instillation site haematoma | 10073609 |
| Instillation site haemorrhage | 10073610 |
| Internal haemorrhage | 10075192 |
| International normalised ratio abnormal | 10022592 |
| International normalised ratio increased | 10022595 |
| Intestinal haematoma | 10069829 |
| Intestinal haemorrhage | 10059175 |
| Intestinal varices haemorrhage | 10078058 |
| Intra-abdominal haematoma | 10056457 |
| Intra-abdominal haemorrhage | 10061249 |
| Intracerebral haematoma evacuation | 10062025 |
| Intracranial haematoma | 10059491 |
| Intracranial tumour haemorrhage | 10022775 |
| Intraocular haematoma | 10071934 |
| Intrapartum haemorrhage | 10067703 |
| Intraventricular haemorrhage | 10022840 |
| Intraventricular haemorrhage neonatal | 10022841 |
| Iris haemorrhage | 10057418 |
| Joint microhaemorrhage | 10077666 |
| Kidney contusion | 10023413 |
| Lacrimal haemorrhage | 10069930 |
| Large intestinal haemorrhage | 10052534 |
| Large intestinal ulcer haemorrhage | 10061262 |
| Laryngeal haematoma | 10070885 |
| Laryngeal haemorrhage | 10065740 |
| Lip haematoma | 10066304 |
| Lip haemorrhage | 10049297 |
| Liver contusion | 10067266 |
| Lower gastrointestinal haemorrhage | 10050953 |
| Lower limb artery perforation | 10075730 |

| MEDDRA Term Name | MEDDRA Code |
|---------------------------------------|-------------|
| Lymph node haemorrhage | 10074270 |
| Mallory-Weiss syndrome | 10026712 |
| Mediastinal haematoma | 10049941 |
| Mediastinal haemorrhage | 10056343 |
| Medical device site bruise | 10075570 |
| Medical device site haematoma | 10075577 |
| Medical device site haemorrhage | 10075578 |
| Melaena | 10027141 |
| Melaena neonatal | 10049777 |
| Meningorrhagia | 10052593 |
| Menometrorrhagia | 10027295 |
| Menorrhagia | 10027313 |
| Mesenteric haematoma | 10071557 |
| Mesenteric haemorrhage | 10060717 |
| Metrorrhagia | 10027514 |
| Mouth haemorrhage | 10028024 |
| Mucocutaneous haemorrhage | 10076048 |
| Mucosal haemorrhage | 10061298 |
| Muscle contusion | 10070757 |
| Muscle haemorrhage | 10028309 |
| Myocardial haemorrhage | 10048849 |
| Myocardial rupture | 10028604 |
| Naevus haemorrhage | 10062955 |
| Nail bed bleeding | 10048891 |
| Nasal septum haematoma | 10075027 |
| Neonatal gastrointestinal haemorrhage | 10074159 |
| Nephritis haemorrhagic | 10029132 |
| Nipple exudate bloody | 10029418 |
| Occult blood positive | 10061880 |
| Ocular retrobulbar haemorrhage | 10057571 |
| Oesophageal haemorrhage | 10030172 |
| Oesophageal intramural haematoma | 10077486 |

| MEDDRA Term Name | MEDDRA Code |
|---------------------------------|-------------|
| Oesophageal ulcer haemorrhage | 10030202 |
| Oesophageal varices haemorrhage | 10030210 |
| Oesophagitis haemorrhagic | 10030219 |
| Optic disc haemorrhage | 10030919 |
| Optic nerve sheath haemorrhage | 10030941 |
| Oral contusion | 10078170 |
| Oral mucosa haematoma | 10074779 |
| Osteorrhagia | 10051937 |
| Ovarian haematoma | 10033263 |
| Ovarian haemorrhage | 10065741 |
| Palpable purpura | 10056872 |
| Pancreatic contusion | 10078654 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatitis haemorrhagic | 10033650 |
| Papillary muscle haemorrhage | 10059164 |
| Paranasal sinus haematoma | 10069702 |
| Parathyroid haemorrhage | 10059051 |
| Parotid gland haemorrhage | 10051166 |
| Pelvic haematoma | 10054974 |
| Pelvic haematoma obstetric | 10034248 |
| Pelvic haemorrhage | 10063678 |
| Penile contusion | 10073352 |
| Penile haematoma | 10070656 |
| Penile haemorrhage | 10034305 |
| Peptic ulcer haemorrhage | 10034344 |
| Pericardial haemorrhage | 10034476 |
| Perineal haematoma | 10034520 |
| Periorbital haematoma | 10034544 |
| Periorbital haemorrhage | 10071697 |
| Periosteal haematoma | 10077341 |
| Peripartum haemorrhage | 10072693 |
| Perirenal haematoma | 10049450 |

| MEDDRA Term Name | MEDDRA Code |
|----------------------------------------------------|-------------|
| Peritoneal haematoma | 10058095 |
| Peritoneal haemorrhage | 10034666 |
| Periventricular haemorrhage neonatal | 10076706 |
| Petechiae | 10034754 |
| Pharyngeal haematoma | 10068121 |
| Pharyngeal haemorrhage | 10034827 |
| Pituitary haemorrhage | 10049760 |
| Placenta praevia haemorrhage | 10035121 |
| Plasminogen activator inhibitor | 10059620 |
| Plasminogen activator inhibitor decreased | 10059619 |
| Plasminogen decreased | 10035493 |
| Plasminogen increased | 10035495 |
| Platelet factor 4 decreased | 10060220 |
| Polymenorrhagia | 10064050 |
| Post abortion haemorrhage | 10036246 |
| Post procedural contusion | 10073353 |
| Post procedural haematoma | 10063188 |
| Post procedural haematuria | 10066225 |
| Post procedural haemorrhage | 10051077 |
| Post transfusion purpura | 10072265 |
| Postmenopausal haemorrhage | 10055870 |
| Postpartum haemorrhage | 10036417 |
| Post-traumatic punctate intraepidermal haemorrhage | 10071639 |
| Procedural haemorrhage | 10071229 |
| Proctitis haemorrhagic | 10036778 |
| Prostatic haemorrhage | 10036960 |
| Protein C increased | 10060230 |
| Protein S abnormal | 10051736 |
| Protein S increased | 10051735 |
| Prothrombin level abnormal | 10037048 |
| Prothrombin level decreased | 10037050 |
| Prothrombin time abnormal | 10037057 |

| MEDDRA Term Name | MEDDRA Code |
|----------------------------------------|-------------|
| Prothrombin time prolonged | 10037063 |
| Prothrombin time ratio abnormal | 10061918 |
| Prothrombin time ratio increased | 10037068 |
| Pulmonary alveolar haemorrhage | 10037313 |
| Pulmonary contusion | 10037370 |
| Pulmonary haematoma | 10054991 |
| Pulmonary haemorrhage | 10037394 |
| Puncture site haemorrhage | 10051101 |
| Purpura | 10037549 |
| Purpura fulminans | 10037556 |
| Purpura neonatal | 10037557 |
| Purpura non-thrombocytopenic | 10057739 |
| Purpura senile | 10037560 |
| Putamen haemorrhage | 10058940 |
| Radiation associated haemorrhage | 10072281 |
| Rectal haemorrhage | 10038063 |
| Rectal ulcer haemorrhage | 10038081 |
| Renal artery perforation | 10075737 |
| Renal cyst haemorrhage | 10059846 |
| Renal haematoma | 10038459 |
| Renal haemorrhage | 10038460 |
| Respiratory tract haemorrhage | 10038727 |
| Respiratory tract haemorrhage neonatal | 10038728 |
| Retinal aneurysm rupture | 10079121 |
| Retinal haemorrhage | 10038867 |
| Retinopathy haemorrhagic | 10051447 |
| Retroperitoneal haematoma | 10058360 |
| Retroperitoneal haemorrhage | 10038980 |
| Retroplacental haematoma | 10054798 |
| Ruptured cerebral aneurysm | 10039330 |
| Russell's viper venom time abnormal | 10059759 |
| Scleral haemorrhage | 10050508 |

| MEDDRA Term Name | MEDDRA Code |
|------------------------------------|-------------|
| Scrotal haematocoele | 10061517 |
| Scrotal haematoma | 10039749 |
| Shock haemorrhagic | 10049771 |
| Skin haemorrhage | 10064265 |
| Skin neoplasm bleeding | 10060712 |
| Skin ulcer haemorrhage | 10050377 |
| Small intestinal haemorrhage | 10052535 |
| Small intestinal ulcer haemorrhage | 10061550 |
| Soft tissue haemorrhage | 10051297 |
| Spermatic cord haemorrhage | 10065742 |
| Spinal cord haematoma | 10076051 |
| Spinal cord haemorrhage | 10048992 |
| Spinal epidural haematoma | 10050162 |
| Spinal epidural haemorrhage | 10049236 |
| Spinal subarachnoid haemorrhage | 10073564 |
| Spinal subdural haematoma | 10050164 |
| Spinal subdural haemorrhage | 10073563 |
| Spleen contusion | 10073533 |
| Splenic artery perforation | 10075738 |
| Splenic haematoma | 10041646 |
| Splenic haemorrhage | 10041647 |
| Splenic varices haemorrhage | 10068662 |
| Splinter haemorrhages | 10041663 |
| Spontaneous haematoma | 10065304 |
| Spontaneous haemorrhage | 10074557 |
| Stoma site haemorrhage | 10074508 |
| Stomatitis haemorrhagic | 10042132 |
| Subarachnoid haematoma | 10076701 |
| Subarachnoid haemorrhage | 10042316 |
| Subarachnoid haemorrhage neonatal | 10042317 |
| Subchorionic haematoma | 10072596 |
| Subchorionic haemorrhage | 10071010 |

| MEDDRA Term Name | MEDDRA Code |
|---------------------------------------------|-------------|
| Subclavian artery perforation | 10075740 |
| Subclavian vein perforation | 10075743 |
| Subcutaneous haematoma | 10042345 |
| Subdural haematoma | 10042361 |
| Subdural haematoma evacuation | 10042363 |
| Subdural haemorrhage | 10042364 |
| Subdural haemorrhage neonatal | 10042365 |
| Subgaleal haematoma | 10069510 |
| Subretinal haematoma | 10071935 |
| Superior vena cava perforation | 10075741 |
| Testicular haemorrhage | 10051877 |
| Thalamus haemorrhage | 10058939 |
| Third stage postpartum haemorrhage | 10043449 |
| Thoracic haemorrhage | 10062744 |
| Thrombin time abnormal | 10051319 |
| Thrombin time prolonged | 10051390 |
| Thrombin-antithrombin III complex abnormal | 10053972 |
| Thrombin-antithrombin III complex increased | 10053968 |
| Thrombocytopenic purpura | 10043561 |
| Thrombotic thrombocytopenic purpura | 10043648 |
| Thyroid haemorrhage | 10064224 |
| Tongue haematoma | 10043959 |
| Tongue haemorrhage | 10049870 |
| Tonsillar haemorrhage | 10057450 |
| Tooth pulp haemorrhage | 10072228 |
| Tooth socket haemorrhage | 10064946 |
| Tracheal haemorrhage | 10062543 |
| Traumatic haematoma | 10044522 |
| Traumatic haemorrhage | 10053476 |
| Traumatic haemothorax | 10074487 |
| Traumatic intracranial haematoma | 10079013 |
| Traumatic intracranial haemorrhage | 10061387 |

| MEDDRA Term Name | MEDDRA Code |
|------------------------------------|-------------|
| Tumour haemorrhage | 10049750 |
| Ulcer haemorrhage | 10061577 |
| Umbilical cord haemorrhage | 10064534 |
| Umbilical haematoma | 10068712 |
| Umbilical haemorrhage | 10045455 |
| Upper gastrointestinal haemorrhage | 10046274 |
| Ureteric haemorrhage | 10065743 |
| Urethral haemorrhage | 10049710 |
| Urinary bladder haemorrhage | 10046528 |
| Urogenital haemorrhage | 10050058 |
| Uterine haematoma | 10063875 |
| Uterine haemorrhage | 10046788 |
| Vaccination site bruising | 10069484 |
| Vaccination site haematoma | 10069472 |
| Vaccination site haemorrhage | 10069475 |
| Vaginal haematoma | 10046909 |
| Vaginal haemorrhage | 10046910 |
| Varicose vein ruptured | 10046999 |
| Vascular access site bruising | 10077767 |
| Vascular access site haematoma | 10077647 |
| Vascular access site haemorrhage | 10077643 |
| Vascular access site rupture | 10077652 |
| Vascular graft haemorrhage | 10077721 |
| Vascular pseudoaneurysm ruptured | 10053949 |
| Vascular purpura | 10047097 |
| Vascular rupture | 10053649 |
| Vein rupture | 10077110 |
| Venous haemorrhage | 10065441 |
| Venous perforation | 10075733 |
| Ventricle rupture | 10047279 |
| Vertebral artery perforation | 10075735 |
| Vessel puncture site bruise | 10063881 |

| MEDDRA Term Name | MEDDRA Code |
|--------------------------------------------|-------------|
| Vessel puncture site haematoma | 10065902 |
| Vessel puncture site haemorrhage | 10054092 |
| Vitreous haematoma | 10071936 |
| Vitreous haemorrhage | 10047655 |
| Von Willebrand's disease | 10047715 |
| Von Willebrand's factor antibody positive | 10066358 |
| Von Willebrand's factor multimers abnormal | 10055165 |
| Vulval haematoma | 10047756 |
| Vulval haematoma evacuation | 10047757 |
| Vulval haemorrhage | 10063816 |
| White nipple sign | 10078438 |
| Withdrawal bleed | 10047998 |
| Wound haematoma | 10071504 |
| Wound haemorrhage | 10051373 |

Appendix 4. List of Medical Search Terms for Diarrhoea

| MEDDRA Term Name | MEDDRA Code |
|-------------------------------------|-------------|
| Defaecation urgency | 10012110 |
| Diarrhoea | 10012735 |
| Diarrhoea haemorrhagic | 10012741 |
| Diarrhoea neonatal | 10012743 |
| Frequent bowel movements | 10017367 |
| Gastrointestinal hypermotility | 10052402 |
| Post procedural diarrhoea | 10057585 |
| Abnormal faeces | 10000133 |
| Allergic gastroenteritis | 10075308 |
| Anal incontinence | 10077605 |
| Antidiarrhoeal supportive care | 10055660 |
| Bowel movement irregularity | 10063541 |
| Change of bowel habit | 10008399 |
| Colitis | 10009887 |
| Colitis erosive | 10058358 |
| Colitis ischaemic | 10009895 |
| Colitis microscopic | 10056979 |
| Colitis psychogenic | 10053397 |
| Culture stool negative | 10011630 |
| Encopresis | 10014643 |
| Enteritis | 10014866 |
| Enteritis leukopenic | 10014877 |
| Enterocolitis | 10014893 |
| Enterocolitis haemorrhagic | 10014896 |
| Eosinophilic colitis | 10057271 |
| Faecal containment device insertion | 10073732 |
| Faecal volume increased | 10049939 |
| Faeces discoloured | 10016100 |
| Gastroenteritis | 10017888 |
| Gastroenteritis eosinophilic | 10017902 |
| Gastroenteritis radiation | 10017912 |
| Gastrointestinal inflammation | 10064147 |

| MEDDRA Term Name | MEDDRA Code |
|------------------------------------|-------------|
| Gastrointestinal motility disorder | 10061173 |
| Gastrointestinal toxicity | 10059024 |
| Gastrointestinal tract irritation | 10070840 |
| Intestinal angioedema | 10076229 |
| Intestinal transit time abnormal | 10074724 |
| Intestinal transit time decreased | 10074598 |
| Irritable bowel syndrome | 10023003 |
| Low anterior resection syndrome | 10080023 |
| Neutropenic colitis | 10062959 |
| Radiation proctitis | 10037766 |